CLINICAL TRIAL: NCT00226200
Title: Soluble CD23 Expression as a Marker of Immunomodulation and CLinical Response in Asthma Patients Treated With Omalizumab
Brief Title: Soluble CD23 Expression in Asthma Patients Treated With OMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Completed
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Gailen D. Marshall. MD, PhD, University of Mississippi Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025AUS10; CIGE025AUS10
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Asthma
Keywords: Allergic; Non allergic
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Omalizumab

SUMMARY:
This study involves a FDA approved drug, Omalizumab, used in the treatment of moderate to severe allergic asthma that cannot be controlled by standard treatment. It works on IgE to control the allergic reaction. We are looking at the effects on non-allergic asthma. We hope to prove that Omalizumab will have the same effect on non-allergic asthmatics as it does allergic asthmatics.

DETAILED DESCRIPTION:
This is a 1 year placebo controlled study looking at moderate to severe asthmatics (allergic or non-allergic) who are controlled by medication.

Skin testing will be done to determine the allergic status, as well as a base line IgE done. The Omalizumab is administered by injection based on weight and IgE level, (once or twice a month).

At several times during the year pulmonary function test will be done, as well blood drawn for immunological assays (CD23 and FcER1 expression, TH1/TH2 cytokines, CD23 production). A battery of questionnaires will also determine quality of life(with asthma), psychological stress measures and parameters of clinical response.

ELIGIBILITY:
Inclusion Criteria:

Moderate to severe asthmatic (based on 1997 NHLBI guidelines), controlled by medication for at least 6 months, initial IgE level between 30 and 700 IU, weigh between 30 an 150 kg, otherwise healthy.

Exclusion Criteria:

Smoker, uncontrolled asthma, immunotherapy in past six weeks, other diseases

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80
Dates: Start 2004-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Measure of sCD23 in plasma
CD23 expression on T cell correlated with spirometry, AQLQ and RQLQ.

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, MD/PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States